CLINICAL TRIAL: NCT02169999
Title: Personalized Decision Support for Older Patients With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 11-0045
Record Dates: First submitted 2014-06-18; First posted 2014-06-23 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Personalized Diabetes Care Website (Experimental): Subjects are exposed to Personalized Diabetes Care website.
  Interventions: Other: Personalized Diabetes Care Website
- No Exposure To Website (No Intervention): Subjects are not exposed to Personalized Diabetes Care website

INTERVENTIONS:
Other: Personalized Diabetes Care Website — Subjects enrolled in the intervention view the Personalized Diabetes Care website and enter their self-reported medical history and personal preferences into the website. A model runs and creates a 2 page print out with risk estimates for the subject to review with their physician.
  Arms: Personalized Diabetes Care Website

SUMMARY:
The purpose of this study is to determine the impact of web-based personalized decision support on:

1. Patient awareness of treatment goal options and ability to articulate their goals of diabetes care.
2. Provider awareness of patients' clinical status (e.g. life expectancy) and treatment preferences.
3. Individualization of care plans in accordance with geriatric diabetes guidelines.

DETAILED DESCRIPTION:
In 2003, the first geriatric diabetes care guidelines were published that encouraged older patients and their providers to consider less intensive glucose control goals (HbA1C <8%) among frail, older patients with limited life expectancy, while continuing to pursue intensive glucose control (HbA1C <7%) among relatively healthy older patients. The guidelines also emphasized the importance of cardiovascular prevention, encouraged routine screening for geriatric syndromes that can influence treatment decisions (i.e., polypharmacy and falls), and advised providers to acknowledge patients' preferences when making treatment decisions.

These guidelines represent a conceptual advance in the care of older diabetes patients; however, there has been little effort to implement and evaluate these recommendations in a practice setting. This may be partially due to the fact that many of the recommendations are difficult to carry out in busy clinical practices without sophisticated decision support tools. Determining whether an older patient will benefit from intensive glucose control is a complex cognitive task requiring simultaneous consideration of multiple, sometimes contradictory, clinical criteria (e.g. advanced duration of diabetes and limited life expectancy). Completing this task accurately may only be possible with computer simulation models.

Along with this barrier to implementing care guidelines, there is also no consensus on how to elicit patient preferences in the setting of chronic disease management or how to account for these views in the decision-making process. To overcome these challenges, we developed a web-based Geriatric Diabetes Decision Aid (GDDA) which combines a decision analytic model of diabetes complications with the latest prognostic tools from geriatrics.

This personalized decision support tool will encourage the individualization of diabetes care among older patients by educating patients on diabetes, delivering prognostic information to providers, providing personalized data on the risks and benefits of diabetes care to patients and providers, and eliciting the treatment preferences of patients. In this proposed set of studies, we developed the GDDA with the input of patients and providers and assessed its impact through individual interviews.

The findings from this series of studies will be important for establishing the feasibility of using the GDDA in practice, and providing estimates of the intervention's effect on processes of care for power calculations for a future large scale randomized controlled trial. This pilot randomized controlled trial will be one of the first trials to formally examine new care recommendations for the growing population of older patients living with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older
* Dx of diabetes
* HbA1C greater than 6.0%
* English speaking

Exclusion Criteria:

* Telephone Mini Mental less than 17
* Blind

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Patients' change in knowledge about diabetes and its treatments | 06/2011 - 12/2013 (32 months)
  We asked patients to identify knowledge of an A1C goal and specific goals for glucose control in pre and post surveys for both arms.

SECONDARY OUTCOMES:
Patients' Change in Decisional Conflict Scores | 6/2011 - 12/2013 (32 months)
  We used the decision conflict scale (10-item) pre and post for both arms to measure any change in patients' decisional conflict regarding choosing their A1C goal.

CONTACTS AND LOCATIONS:
Overall Officials: Elbert S Huang, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Hospitals, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang ES, Nathan AG, Cooper JM, Lee SM, Shin N, John PM, Dale W, Col NF, Meltzer DO, Chin MH. Impact and Feasibility of Personalized Decision Support for Older Patients with Diabetes: A Pilot Randomized Trial. Med Decis Making. 2017 Jul;37(5):611-617. doi: 10.1177/0272989X16654142. Epub 2016 Jun 16. PMID 27311651